CLINICAL TRIAL: NCT06858995
Title: Experience of PLUVICTO (PSMA-617 Labelled With Lutetium-177) Administration on Totally Implantable Venous Access Port (TIVAP)
Brief Title: Experience of 177Lu-PSMA-617-administration on Port Reservoir (TIVAP)
Acronym: PLUVIPAC
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BOURSIER Caroline, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2025PI037
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Administration of Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: to measure the residual activity on the Totally Implantable Venous Access Port — VOI (volume of interest)TIVAP at 4 ml were drawn manually on the chamber of the TIVAP on each tomography. Blood background was determined by an VOI (volume of intesrest of Right Auricle on the right atrium. The VOIRA was automatically delineated on the CT by XXX. Standardized Uptake Value (SUV)max, SUVpeak, SUVmean were extracted from the VOIs and unilateral comparisons of superiority were performed using Wilcoxon tests. A qualitative analysis along the (TIVAP) catheter was performed: positive if an uptake was superior to the blood background and negative if any.

SUMMARY:
According to Pluvicto® indication, most of patients treated are elderly, with limited/poor venous peripheric access but they received previously chemotherapy through TIVAP and TIVAP generally stays in the body of patients when they are referred for Pluvicto® therapy. This is why TIVAP could be an interesting alternative for administering of 177Lu-PSMA-617. The aim of this study is to assess potential retention of 177Lu-PSMA-617 on TIVAP during administration through in vitro/ex vivo experimentations then in in vivo analysis.

DETAILED DESCRIPTION:
Pluvicto® (177Lu-PSMA-617) was approved in the USA by the Food and Drug Administration (FDA) in March 2022 and in Europe in December 2022 for the treatment of adult patients with progressive, prostate-specific membrane antigen (PSMA)-positive, castration-resistant, metastatic prostate cancer (mCRPC) who have been treated with androgen pathway-inhibiting hormone therapy and taxane-based chemotherapy. The European Medicines Agency (EMA) and FDA recommends using an intravenous catheter exclusively for Pluvicto® administration, which implies that Pluvicto® administration has not to be administreted into a Totally Implantable Venous Access Port (TIVAP). In fact, administration through central venous access is preferred for repeated venous infusion in particular in oncology patients for preventing damage veins, and painful and TIVAPs is particular used for intensive and long-term chemotherapy in most oncology departments. However, according to Pluvicto® indication, most of patients treated are elderly, with limited/poor venous peripheric access but they received previously chemotherapy through TIVAP and TIVAP generally stays in the body of patients when they are referred for Pluvicto® therapy. This is why TIVAP could be an interesting alternative for administering of 177Lu-PSMA-617. The aim of this study is to assess potential retention of 177Lu-PSMA-617 on TIVAP during administration through in vitro/ex vivo experimentations then in in vivo analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an injection of Pluvicto as part of the treatment of their prostate cancer, having had a SPECT/CT scan for dosimetry within 2 to 4 hours after injection.

Exclusion Criteria:

* Patients who have refused to have their data used for research purposes

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients following an injection of Pluvicto as part of the treatment of their prostate cancer, having had a SPECT/CT scan for dosimetry within 2 to 4 hours after injection over the period from February 2022 to October 2023 are concerned by this study.
Sampling Method: Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Show that the residual activity at the port reservoir level is negligible, there is no 177Lu-PSMA-617 accumulation at the port reservoir level above the blood background noise | 1 day
  The 4 ml regions of interest (VOI = volume of interest) were manually drawn on the PAC on each SPECT/CT. The blood background was determined by a VOI drawn on the right atrium

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de NANCY, Vandœuvre-lès-Nancy
  - Nuclear medicine Department CHRU de NANCY, Vandœuvre-lès-Nancy